CLINICAL TRIAL: NCT06040359
Title: Pilot Evaluation of the Thriving Mamas Programme for Adolescent Perinatal Mental Health
Brief Title: Pilot Evaluation of the Thriving Mamas Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Aga Khan University (Other); Centro Internacional para Saude Reprodutiva Mocambique (Unknown); UK Research and Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HR/DP-22/23-39521
Record Dates: First submitted 2023-08-23; First posted 2023-09-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Perinatal Mental Health
Keywords: Adolescent mental health; Maternal mental health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thriving Mama programme (Experimental): Nine meetings delivered in either group (5 meetings), individual (1 meeting), or family group (2 meetings) formats over 10 weeks with an additional individual meeting 10-12 weeks postpartum by a trained mother in the community. Each meeting focuses on the girl's physical and mental health, taking care of a newborn, life skills, future-planning and social support and community-based services. Meetings will take place in a mixture of private settings in health facilities, community facilities, and participant homes. Adolescents will also receive usual perinatal care.
  Interventions: Other: The Thriving Mamas programme
- Usual perinatal care (Active Comparator): Each visit includes care that is appropriate to the overall condition and stage of pregnancy and should include four main categories of care:
  1. Identification of pre-existing health conditions (e.g., check for weight and nutrition status, anemia, hypertension, syphilis, HIV status);
  2. Early detection of complications arising during pregnancy (e.g., check for pre-eclampsia, gestational diabetes);
  3. Health promotion and disease prevention (e.g., tetanus vaccine, prevention and treatment of malaria, nutrition counseling, micronutrient supplements, family planning counseling); and
  4. Birth preparedness and complication planning (e.g., birth and emergency plan, breastfeeding counseling, antiretrovirals for HIV positive women and reducing mother-to- child transmission of HIV)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: The Thriving Mamas programme — Enhanced antenatal course plus usual perinatal care
  Arms: Thriving Mama programme
Other: Usual care — Usual perinatal care
  Arms: Usual perinatal care

SUMMARY:
The goal of this pilot study is to evaluate the feasibility, appropriateness, and acceptability of a mental health prevention intervention among adolescents during pregnancy and the year after birth (perinatal period) in Kenya and Mozambique. The main questions it aims to answer are:

* Is the intervention feasible, acceptable, appropriate, and delivered/received with high fidelity, to adolescent girls, their friends/family members and service providers?
* Are the implementation strategies acceptable, appropriate, feasible to all relevant stakeholders?
* What impact does the intervention have on adolescent mothers' mental health?
* What impact does the intervention have on adolescent mothers' social, economic, and education outcomes?

Participants will:

* Participate in nine individual and group sessions focused on improving mental and perinatal health literacy and increasing life skills
* Receive standard perinatal care

Researchers will compare findings with girls receiving standard perinatal care only to see if the intervention has an impact on adolescents' mental health, social, economic and education outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Mentor mothers: (A) aged 20 years or older; (B) female; (C) experience of pregnancy and/or parenting; and (D) live within the study site
* Adolescent girls: (A) up to 28 weeks pregnant; and (B) aged 15-19 years
* Friends/family members: (A) identified by an adolescent or young woman participating in the study; (B) participation agreed by other participating girls; and (C) aged 18 years or older

Exclusion Criteria:

* Mentor mothers will be excluded from participating if they are unable to attend training or deliver the intervention sessions
* Adolescent girls will be excluded from the study if they are unable to provide informed consent or are unable to participate in the intervention, due to existing health conditions
* Friends/family members will not be excluded so long as they meet inclusion criteria

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 10-12 weeks post-partum
  Feasibility of Intervention Measure (FIM); Subjective report of feasibility of intervention; measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Minimum=5, Maximum=25; higher score is better
Intervention Acceptability | 10-12 weeks post-partum
  Acceptability of Intervention Measure (AIM); Subjective report of acceptability of intervention; A 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Minimum=5, Maximum=25; higher score is better
Intervention Appropriateness | 10-12 weeks post-partum
  Intervention Appropriateness Measure (IAM); Subjective report of appropriateness of intervention; A 5-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. Minimum=5, Maximum=25; higher score is better
Intervention Fidelity | Through intervention delivery, an average of 24 weeks
  Enhancing Assessment of Common Therapeutic Factors (ENACT); subjective report of provider fidelity and perception of care; Minimum=0; Maximum=13; higher score is better

SECONDARY OUTCOMES:
Training Feasibility | Immediately after provider training
  Feasibility of Intervention Measure (FIM); Subjective report of feasibility of intervention; measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Minimum=5, Maximum=25; higher score is better
Training Acceptability | Immediately after provider training
  Acceptability of Intervention Measure (AIM); Subjective report of acceptability of intervention; A 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Minimum=5, Maximum=25; higher score is better
Training Appropriateness | Immediately after provider training
  Intervention Appropriateness Measure (IAM); Subjective report of appropriateness of intervention; A 5-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. Minimum=5, Maximum=25; higher score is better
Knowledge | Baseline and immediately after provider training
  Study-specific measure of mentor mothers' knowledge of issues regarding pregnancy, childbirth, caregiving, mental health, and referral pathways will be assessed using a study-specific quiz based upon the intervention manual; Minimum=0, Maximum=16; higher score is better
Change in mental health attitudes | Baseline and immediately after provider training
  Social Distance Scale (SDS); The SDS measures the acceptability of different degrees of social distance and, by inference, the attitude of the respondent to the person with the condition; Minimum=1, Maximum=96; higher score is better
Change in adolescent pregnancy attitudes | Baseline and immediately after provider training
  Study-specific attitudes towards adolescent pregnancy survey; Minimum=4, Maximum=20; lower score is better
Provider competency | Immediately after provider training
  Study-specific single 10-point scale to assess provider ability to deliver the intervention; Minimum=0, Maximum=10; higher score is better
Recruitment rate | pre-intervention
  Proportion of adolescents providing consent to participate in the study
Cost of intervention | through study completion, an average of 24 weeks
  Total and average cost of the intervention per participant
Change in adolescent depression | through study completion, an average of 24 weeks
  Patient Health Questionnaire (PHQ-9); Nine-item screening tool which assesses depression symptoms according to clinical criteria. Minimum=0, Maximum=27. A score ≥10 indicates moderate to severe depression.
Change in adolescent anxiety | through study completion, an average of 24 weeks
  Generalised Anxiety Disorder scale (GAD-7); Seven-item screening tool which assesses anxiety symptoms according to clinical criteria. Minimum=0, Maximum=21. A score ≥10 indicates moderate to severe anxiety.
Change in adolescent quality of life | through study completion, an average of 24 weeks
  WHO Quality of Life brief version (WHOQOL-BREF); 26-item scale assesses a respondent's perceived quality of life across four domains: physical health; psychological; social relationships; and environment. Total minimum=25, Total maximum=125. Higher scores indicate greater quality of life in a particular domain.
Change in adolescent social support | through study completion, an average of 24 weeks
  Multidimensional Scale of Perceived Social Support (MSPSS); The MSPSS is a 12-item scale which measures social support from family, friends and significant others. Minimum=12, Maximum=84. Higher scores indicate greater social support.
Adolescent parenting competency | through study completion, an average of 24 weeks
  Parenting Sense of Competency Scale; 17-item scale to measure adolescents' perceived parenting abilities. Minimum=17, Maximum=102. Higher scores indicate greater perceived competence.
Perinatal appointment attendance | through study completion, an average of 24 weeks
  Number of participants attending antenatal appointments
Referral uptake | 10-12 weeks post-partum
  Proportion of adolescents attending referral appointments
Change in infant vaccination | Baseline and 10-12 weeks post-partum
  Number of participants intending to or having had their babies vaccinated
Change in breastfeeding | Baseline and 10-12 weeks post-partum
  Number of participants intendng to or are currently breastfeeding
Change in intended time to next pregnancy | Baseline and 10-12 weeks post-partum
  Study-specific health behaviours questionnaire to assess intended or actual contraceptive Nuimber of participants that want more children who intend to wait at least 15 months before next pregnancy
Change in contraceptive use | Baseline and 10-12 weeks post-partum
  Number of participants intending to or currently using contraceptives to delay pregnancy
Change in perception of intervention | Baseline and 10-12 weeks post-partum
  Study-specific five-item measure assessing knowledge gained, interest in intervention, and support recieved; Minimum=0; Maximum=5; higher score is better

CONTACTS AND LOCATIONS:
Locations (2):
- Aga Khan University, Nairobi, Kenya
- Centro Internacional para Saude Reprodutiva Mocambique, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Taylor Salisbury T, Maguele MSB, Chissale F, de Melo M, Hanselmann M, Lamahewa K, Lang'at E, Mandlate F, Nyaga L, Seward N, Temmerman M. Supporting the mental health of adolescent mothers in Kenya and Mozambique: pilot protocol for the Thriving Mamas programme. Pilot Feasibility Stud. 2025 Jun 19;11(1):83. doi: 10.1186/s40814-025-01617-5. PMID 40537871